CLINICAL TRIAL: NCT02797119
Title: Tranexamic Acid to Reduce Blood Loss in Hemorrhagic Caesarean Delivery: a Multicenter Randomized Double Blind Placebo Controlled Therapeutic and Pharmaco-biological Dose Ranging Study (TRACES) for Its Optimal Benefit/Risk
Brief Title: Tranexamic Acid to Reduce Blood Loss in Hemorrhagic Caesarean Delivery
Acronym: TRACES
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study will be stopped due to the impossibility of reaching the objective of inclusions within a reasonable time frame and taking into account the recommendations of the international WOMAN study
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government); French Health Products Safety Agency (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015_13; 2015-002499-26 (EudraCT Number); PHRC_2014_0032 (Other: PHRC number, DGOS)
Record Dates: First submitted 2016-05-17; First posted 2016-06-13 (Estimated); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Pregnancy Complications; Hemorrhage
Keywords: Tranexamic acid; Fibrinolysis; Cesarean section; Pharmacokinetics; D dimers; Fibrinogen; Plasmin; Transfusion
MeSH Terms: conditions — Pregnancy Complications; Hemorrhage | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- tranexamic acid 1 g (TA1) (Experimental): To measure the efficacy of a standard 1g dose TA to reduce blood loss in ongoing hemorrhagic cesarean section.
  To correlate this clinical effect with the fibrinolysis inhibition and the TA venous and uterine blood concentration
  Interventions: Drug: tranexamic acid 1 g (TA1)
- tranexamic acid 0.5 g (TA1/2) (Experimental): To measure the efficacy of a low 0,5g dose TA to reduce blood loss in ongoing hemorrhagic cesarean section To correlate this clinical effect with the fibrinolysis inhibition and the TA venous and uterine blood concentration
  Interventions: Drug: tranexamic acid 0.5 g (TA1/2)
- Saline Solution (TA0) (Placebo Comparator): To measure the evolution of blood loss without TA in ongoing hemorrhagic cesarean section To correlate this clinical evolution with fibrinolysis.
  Interventions: Drug: Saline Solution (TA0)
- NH (No Intervention): To measure the reference fibrinolytic activity in non-hemorrhagic cesarean section

INTERVENTIONS:
Drug: tranexamic acid 1 g (TA1) — 1 g standard dose tranexamic acid, intravenous unique bolus over 1 minute
  Arms: tranexamic acid 1 g (TA1)
Drug: tranexamic acid 0.5 g (TA1/2) — 0.5 g standard dose tranexamic acid, intravenous unique bolus over 1 minute
  Arms: tranexamic acid 0.5 g (TA1/2)
Drug: Saline Solution (TA0)
  Arms: Saline Solution (TA0)

SUMMARY:
TRACES trial is a multicenter randomized double blind placebo control therapeutic and pharmaco-biological dose ranging study to measure the effect on blood loss reduction of a single intravenous infusion of two doses regimens (standard dose and low dose) of TA administered at the onset of an active PPH (>800mL) during elective or non-emergent CS and to correlate this clinical effect with the biological effect of fibrinolysis inhibition and the pharmacodynamic measure of TA uterine bleeding and venous blood concentration.

DETAILED DESCRIPTION:
Postpartum hemorrhage (PPH) is the leading cause of maternal death. Tranexamic acid (TA) (Exacyl® Sanofi France), an antifibrinolytic drug, reduces bleeding and transfusion need in major surgery and trauma (1). In ongoing PPH following vaginal delivery (2), a high dose of TA decreased the volume and duration of PPH, the transfusion need and the maternal morbidity, while early fibrinolysis was inhibited (3). Prophylactic use of TA limited the postoperative bleeding in elective non hemorrhagic caesarean section (CS). (1, 4) TA efficiency in the hemorrhagic caesarean context has not been previously published.

TA doses range vary from 2,5 to 100 mg/kg and side effects were observed with the largest doses.(1,4) Pharmacokinetics old data concerned non hemorrhagic patients.(1) WOMAN ongoing international trial using a one gram dose have a mortality reduction objective.(5) The optimal dose for ongoing caesarean PPH has to be determined.

Aim of the study:

The aim of the multicenter randomized double blind placebo control therapeutic and pharmaco-biological dose ranging study TRACES is to measure the effect on blood loss reduction of a single intravenous infusion of two doses regimens of TA administered at the onset of an active PPH (>800mL) during elective or non-emergent CS and to correlate this clinical effect with the biological effect of fibrinolysis inhibition and the pharmacodynamic measure of TA uterine bleeding and venous blood concentration.

Statistical method:

The sample size computation is based on the expected difference between the placebo group and the low dose. On the base of EXADELI trial results, the investigators calculated that a total of 342 subjects (114 per group) is required, For the main objective, the blood loss volume measured in each experimental group (low dose and high dose) will be compared to that of the placebo group by using an analysis of covariance adjusted for baseline blood loss volume. In cases of non-normal distribution, relative blood loss volume will be calculated and compared using a Mann-Whitney U test. Analyses will be done on an intention-to-treat basis and all statistical tests will be performed with a 2-tailed alpha risk of 0.05. The sample size computation for the pharmaco-biological substudy have been calculated regarding the inhibition of fibrinolysis (D Dimers increase between 30 and 120 minutes negative or null (EXADELI trial 11)). The NNS for this substudy is 48 patients in each of the 3 hemorrhagic groups and 48 patients in the reference non-hemorrhagic group for a total of 192 patients. These substudy hemorrhagic patients will be selected from the experimental groups as the first 144 patients for which the TA concentration and plasmin peak specific sampling will be completed regarding the blood collection and congelation organisation in each center.

Expected research benefit:

The project is aimed to answer for a current clinical practice question: Timing and dose of TA to reduce blood loss and maternal morbidity due to active hemorrhage during CS in order to determine the optimal and minimal TA dose to obtain the better efficacy and the limitations of side-effects.

ELIGIBILITY:
Inclusion Criteria:

Experimental group: Each patient

* experiencing a bleeding volume of more than 800 mL
* due to surgery or to atony uterine
* during an elective or non-emergent caesarean section
* secondary post-partum haemorrhage after caesarean section, even if CS has been emergent
* after complete information and consent signature.
* covered by social security. Reference non-hemorrhagic group: Each patient
* experiencing a bleeding volume of strictly less than 800 mL
* during an elective or emergent caesarean section
* after complete information and consent signature.
* covered by social security.

Exclusion Criteria:

Patient unable to consent (<18 years old or incapable people and specially protected mentioned in the article L1121-5 to L1121-8) RCP medical contraindication to tranexamic acid such as

* Hypersensibility to the product or excipient,
* Previous or ongoing arterial or venous thrombosis,
* Coagulopathy, except DIC associated with a predominant fibrinolytic profile,
* Renal failure,
* Previous seizures,
* intrathecal or intraventricular administration. Obstetrical contraindication to TA
* Severe HELLP syndrome (platelet count <50 000/m3 or renal failure prior to the caesarean (RIFLE score>2) Protocol related contraindication to inclusion
* Administration of TA before inclusion-Inherited haemorrhagic diseases and low molecular weight heparin within 24 hours before inclusion
* Patients who participated in a study on the efficacy of an experimental drug in the two month preceding the caesarean section
* Inherited haemorrhagic diseases or low molecular weight heparin within 24 hours before inclusion
* Previous inclusion in an interventional trial since the 2 months before CS

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 225 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Bleeding | between inclusion (T0) and 6 hours after inclusion (T360).
  Bleeding will be strictly measured (mL) in aspiration or cell salvage bags (substraction of the amniotic fluid if needed) and drapes weighting at each time point.

SECONDARY OUTCOMES:
Postpartum anemia | at day 2, at day 5
Postpartum blood loss | at Day 2
number of patients presenting with maternal morbidity ie haemostatic interventions and organ failure and ICU admission | At day 5, At day 42
Death | at day 42
Biological fibrinolysis inhibition | Between T0 (inclusion) and T360 (6hours later)
  Percentage of patients for which D Dimers increase is blunted.
Urinary urea and Creatinuria on timed diuresis | Between T0 (inclusion) and T360 (6hours later)
  Urinary Urea (g/L) and creatinuria (mg/L) are measured on a timed urinary sample : collected from the bladder catheter, initial diuresis at the beginning of CS is thrown out at the time of inclusion. A strict measure of urinary volume is made at T120, a sample of one monovette of urines is done to get the concentration of urea, creatinuria and tranexamic acid and their ratio and then thrown out. The same process is done on the urinary volume collected between T120 and T360.
the number of patients developing an oliguria or a renal failure (RIFLE score more than 2) | Between T0 (inclusion) and T360 (6hours later)
  Diuresis is measured on a timed urinary sample : collected from the bladder catheter, initial diuresis at the beginning of CS is thrown out at the time of inclusion. A strict measure of urinary volume is made at T120 and T360. Oliguria is defined as a diuresis less than 180mL per 6 hours. Urea (g/L) and creatininemia (mg/L) are measured at T0 inclusion and T360, 6 hours later. the number of patients developping an oliguria or a renal failure (RIFLE score more than 2) is collected.
Deep vein thrombosis or pulmonary embolism | Between T0 (inclusion) and Day 42
  Number of patient developing a deep vein thrombosis or pulmonary embolism clinically diagnosed and confirmed by echodoppler for DVT and angiosccanner for PE. Data collected from the clinical follow up since hospital discharge and a phone call at D42 +/- 10 days
Seizures | Between T0 (inclusion) and Day 42
  Number of patient developing a seizure clinically diagnosed
Visual disturbances | Between T0 (inclusion) and Day 42
  Number of patient developing a colours' visual disturbance clinically diagnosed. Data collected from the clinical follow up since hospital discharge and a phone call at D42 +/- 10 days.
Nausea | Between T0 (inclusion) and Day 42
  Number of patient developing nausea clinically diagnosed and needing a treatment. Data collected from the clinical follow up since hospital discharge and a phone call at D42 +/- 10 days.
Peak Plasma Concentration (Cmax) in venous blood | Between T0 (inclusion) and T360 (6hours after inclusion)
  Venous blood sampled on a dedicated catheter. Biological assessment using Van Geffen method for thrombin and plasmin direct measurement in a weill. Plasmin inhibition.
Area under the plasma concentration versus time curve (AUC) in venous blood | Between T0 (inclusion) and T360 (6hours after inclusion)
  Venous blood sampled on a dedicated catheter. Biological assessment using Van Geffen method for thrombin and plasmin direct measurement in a weill.
Lagtime between thrombin and plasmin peaks (s) in venous blood | Between T0 (inclusion) and T360 (6hours after inclusion)
  Venous blood sampled on a dedicated catheter. Biological assessment using Van Geffen method for thrombin and plasmin direct measurement in a weill.
Peak Plasma Concentration (Cmax) in uterine bleeding | Between T0 (inclusion) and T360 (6hours after inclusion)
  Uterine bleeding sampled by obstetrician in placental bed and after hysterotomy is closed, collected vaginally. Biological assessment using Van Geffen method for thrombin and plasmin direct measurement in a weill.
Area under the plasma concentration versus time curve (AUC) in uterine bleeding | Between T0 (inclusion) and T360 (6hours after inclusion)
  Uterine bleeding sampled by obstetrician in placental bed and after hysterotomy is closed, collected vaginally. Biological assessment using Van Geffen method for thrombin and plasmin direct measurement in a weill.
Lagtime between thrombin and plasmin peaks (s) in uterine bleeding | Between T0 (inclusion) and T360 (6hours after inclusion)
  Uterine bleeding sampled by obstetrician in placental bed and after hysterotomy is closed, collected vaginally. Biological assessment using Van Geffen method for thrombin and plasmin direct measurement in a weill.
Tranexamic acid plasma concentration | Between T0 (inclusion) and T360 (6hours after inclusion)
  Venous blood sampled on a dedicated catheter. Biological assessment using direct plasma drug concentration (mg/L) measurement.
Tranexamic acid concentration in uterine bleeding | Between T0 (inclusion) and T360 (6hours after inclusion)
  Uterine bleeding sampled by obstetrician in placental bed and after hysterotomy is closed, collected vaginally. Biological assessment using direct plasma drug concentration (mg/L) measurement.
Tranexamic acid urinary excretion | Between T0 (inclusion) and T360 (6hours after inclusion)
  Tranexamic acid concentration (mg/L) is measured parallely to urinary urea (g/L) and creatinuria (mg/L) on a timed urinary sample : collected from the bladder catheter, initial diuresis at the beginning of CS is thrown out at the time of inclusion. A strict measure of urinary volume is made at T120, a sample of one monovette of urines is done to get the concentration of urea, creatinuria and tranexamic acid and their ratio and then thrown out. The same process is done on the urinary volume collected between T120 and T360.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie Ducloy-Bouthors, MD, Principal Investigator — University Hospital, Lille
Locations (5):
- France (5):
  - Hôpital Jeanne de Flandre - CHRU de Lille, Lille
  - Hospices civils de Lyon CHU-Lyon Croix Rousse, Lyon
  - Assistance Publique Hôpitaux Paris Hôpital Louis Mourier, Paris
  - Assistance Publique Hôpitaux Paris Hôpital Trousseau, Paris
  - Centre Hospitalier Maternité Monaco Valenciennes, Valenciennes

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van Geffen M, Loof A, Lap P, Boezeman J, Laros-van Gorkom BA, Brons P, Verbruggen B, van Kraaij M, van Heerde WL. A novel hemostasis assay for the simultaneous measurement of coagulation and fibrinolysis. Hematology. 2011 Nov;16(6):327-36. doi: 10.1179/102453311X13085644680348. PMID 22183066
- [Result] Ducloy-Bouthors AS, Jude B, Duhamel A, Broisin F, Huissoud C, Keita-Meyer H, Mandelbrot L, Tillouche N, Fontaine S, Le Goueff F, Depret-Mosser S, Vallet B; EXADELI Study Group; Susen S. High-dose tranexamic acid reduces blood loss in postpartum haemorrhage. Crit Care. 2011;15(2):R117. doi: 10.1186/cc10143. Epub 2011 Apr 15. PMID 21496253
- [Result] Anne-Sophie Ducloy-Bouthors, Alain Duhamel, Antoine Tournoys, Annabelle, Gisele Debize, Edith Peneau, Brigitte Jude, Benoit Vallet, Dominique De Prost, Cyril Huissoud, Sophie Susen., Hyperfibrinolysis and post-partum haemorrhage induced coagulopathy. 2013, Thrombosis research Volume 131, Supplement S88-89. Accepted BJA-2014-00923.
- [Result] Goobie SM, Meier PM, Sethna NF, Soriano SG, Zurakowski D, Samant S, Pereira LM. Population pharmacokinetics of tranexamic acid in paediatric patients undergoing craniosynostosis surgery. Clin Pharmacokinet. 2013 Apr;52(4):267-76. doi: 10.1007/s40262-013-0033-1. PMID 23371895
- [Result] Rozen L, Faraoni D, Sanchez Torres C, Willems A, Noubouossie DC, Barglazan D, Van der Linden P, Demulder A. Effective tranexamic acid concentration for 95% inhibition of tissue-type plasminogen activator induced hyperfibrinolysis in children with congenital heart disease: A prospective, controlled, in-vitro study. Eur J Anaesthesiol. 2015 Dec;32(12):844-50. doi: 10.1097/EJA.0000000000000316. PMID 26258658
- [Derived] Ducloy-Bouthors AS, Gilliot S, Kyheng M, Faraoni D, Turbelin A, Keita-Meyer H, Rigouzzo A, Moyanotidou G, Constant B, Broisin F, Gouez AL, Favier R, Peynaud E, Ghesquiere L, Lebuffe G, Duhamel A, Allorge D, Susen S, Hennart B, Jeanpierre E, Odou P; TRACES working group. Tranexamic acid dose-response relationship for antifibrinolysis in postpartum haemorrhage during Caesarean delivery: TRACES, a double-blind, placebo-controlled, multicentre, dose-ranging biomarker study. Br J Anaesth. 2022 Dec;129(6):937-945. doi: 10.1016/j.bja.2022.08.033. Epub 2022 Oct 13. PMID 36243576
- [Derived] Ducloy-Bouthors AS, Jeanpierre E, Saidi I, Baptiste AS, Simon E, Lannoy D, Duhamel A, Allorge D, Susen S, Hennart B. TRAnexamic acid in hemorrhagic CESarean section (TRACES) randomized placebo controlled dose-ranging pharmacobiological ancillary trial: study protocol for a randomized controlled trial. Trials. 2018 Mar 1;19(1):149. doi: 10.1186/s13063-017-2421-6. PMID 29490690
- [Derived] Bouthors AS, Hennart B, Jeanpierre E, Baptiste AS, Saidi I, Simon E, Lannoy D, Duhamel A, Allorge D, Susen S. Therapeutic and pharmaco-biological, dose-ranging multicentre trial to determine the optimal dose of TRAnexamic acid to reduce blood loss in haemorrhagic CESarean delivery (TRACES): study protocol for a randomised, double-blind, placebo-controlled trial. Trials. 2018 Mar 1;19(1):148. doi: 10.1186/s13063-017-2420-7. PMID 29490682